CLINICAL TRIAL: NCT03235960
Title: Clinical Efficacy of Glass-ionomer Fissure Sealants
Brief Title: Efficacy of Glass-ionomer Fissure Sealants
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Association of Paediatric and Preventive Dentists of Serbia (Other)
Responsible Party: Principal Investigator, Dejan Markovic, professor, Association of Paediatric and Preventive Dentists of Serbia
Other Study IDs: 001-04
Record Dates: First submitted 2017-07-18; First posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-07

CONDITIONS: Fissure Sealant; Glass-ionomer Cement; Permanent Molar

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: glass-ionomer fissure sealant — The encapsulated glass-ionomer cement for fissure protection was applied onto the selected permanent molar according to the manufacturer's instruction

SUMMARY:
Despite numerous techniques for enamel protection, occlusal caries still remains a problem. Sealing pits and fissures is considered to be an effective way of preventing caries development. Glass-ionomer cements are mainly recommended for pits and fissures sealing for two reasons. First, they are less susceptible to moisture which allows their use in noncooperable children or in partially erupted teeth where isolation could be a problem, and secondly, due to their potential to act as a fluoride reservoir making enamel more resistant to demineralisation. The purpose of the study is to clinically examine the caries-preventive effect of a glass-ionomer material for fissure protection in newly erupted permanent molars in children with low, moderate, and high caries-risk.

DETAILED DESCRIPTION:
Despite numerous techniques for enamel protection, such as topical fluorides, calcium phosphate-based remineralization systems, xylitol, etc., occlusal caries still remains a problem. A carious lesion occurs in pits and fissures of occlusal surfaces primarily due to their specific anatomy, which is considered to be an ideal site for the retention of bacteria and food remnants rendering mechanical means of debridement inaccessible. Sealing pits and fissures is considered to be an effective way of preventing caries development. Today, there is a wide spectrum of available sealing materials. Glass-ionomer cements are mainly recommended for pits and fissures sealing for two reasons. First, they are less susceptible to moisture which allows their use in noncooperable children or in partially erupted teeth where isolation could be a problem, and secondly, due to their potential to act as a fluoride reservoir making enamel more resistant to demineralisation. During last decades, glass-ionomer cements of different physical and chemical properties were used for pits and fissure sealing which probably contributed to variances in their clinical efficacy. The purpose of the study is to clinically examine the caries-preventive effect of a glass-ionomer material for fissure protection in newly erupted permanent molars in children with low, moderate, and high caries-risk.

ELIGIBILITY:
Inclusion Criteria:

* at least one recently erupted permanent molar with sound pits and fissures
* healthy patients
* possibility to perform a dental treatment
* willing to participate in the study

Exclusion Criteria:

* teeth with an obvious cavity, with a restoration or a sealant completely or partially presented in the fissure system
* medically compromised patients
* non cooperative patients
* not willing to participate in the study

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Healthy children who appeared for a regular dental examination
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2004-01-01 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-08-01 (Estimated)

PRIMARY OUTCOMES:
absence of caries | every 12 months during 13 years
  absence of caries on sealed tooth surfaces
retention of sealant | every 12 months during 13 years
  complete or partial retention

CONTACTS AND LOCATIONS:
Overall Officials: Dejan Markovic, PhD, Principal Investigator — University of Belgrade, School of Dental Medicine
Locations (1):
- University of Belgrade, School of Dental Medicine, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: No